CLINICAL TRIAL: NCT06457373
Title: The Demineralized Dentin Allograft Versus Demineralized Dentin Autograft for Socket Preservation After Surgical Extraction of Impacted Mandibular Third Molar
Brief Title: Demineralized Dentin Allograft Versus Demineralized Dentin Autograft for Socket Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Habib, Oral and maxillofacial surgery clinical demonstrator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (DDA) for socket preservation
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Bone Loss
Keywords: Socket preservation; Impacted mandibular third molar; Alveolar ridge Augmentation
MeSH Terms: conditions — Alveolar Bone Loss | interventions — bis(p-chlorophenyl)acetic acid

STUDY DESIGN:
Intervention Model Description: 20 sockets will be grafted with Demineralized Dentin Allograft (DDA) and 20 sockets will be grafted with Demineralized Dentin Autograft (Auto-DD)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 20 sockets will be grafted with Demineralized Dentin Allograft (DDA)
  Interventions: Procedure: Demineralized Dentin Allograft
- Group B (Active Comparator): 20 sockets will be grafted with Demineralized Dentin Autograft (Auto-DD)
  Interventions: Procedure: Demineralized Dentin Autograft

INTERVENTIONS:
Procedure: Demineralized Dentin Allograft — 20 sockets are randomly allocated to receive the Demineralized Dentin Allograft (split-mouth study)
  Other Names: DDA
  Arms: Group A
Procedure: Demineralized Dentin Autograft — 20 sockets are randomly allocated to receive the Demineralized Dentin Autograft (split-mouth study)
  Other Names: Auto-DD
  Arms: Group B

SUMMARY:
This study is designed to evaluate and compare clinically and radiographically the effectiveness of Demineralized Dentin Allograft (DDA) versus Demineralized Dentin Autograft (Auto-DD) for preservation of alveolar ridge dimensions after surgical extraction of the impacted mandibular third molar.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 25 to 35 years old.
2. Patients scored as (ASA I).
3. No adverse habits such as smoking, tobacco chewing, alcohol.
4. Patients having bilaterally impacted mandibular third molar with similar degree of difficulty according to (Kim JY, et al).
5. The recipient alveolar sockets are free of any pre-existing periapical pathology, based on x-ray.
6. Alveolar sockets with a depth of 5 mm or more, using periodontal probe for assessment.
7. Patients sign a consent for all procedures.

Exclusion Criteria:

* 1) Pregnant or lactating patients. 2) Relevant systemic diseases. 3) Patients with history of chemotherapy or radiotherapy.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Measuring and comparing the height of bone between the two groups | Immediately post-operative, 3months post-operative, 6months post-operative
  We will measure the height of the alveolar ridge clinically by using ridge mapping caliper (special caliper forceps used for measuring ridge dimensions) and radiographically on the cone-beam computed tomography (CBCT) and comparing the results of the study group (20 sockets) with the control group (the other 20sockets), to assess the effectiveness of Demineralized Dentin Allograft for ridge preservation
Measuring and comparing the width of bone between the two groups | Immediately post-operative, 3months post-operative, 6months post-operative
  We will measure the width of the alveolar ridge clinically by using ridge mapping caliper (special caliper forceps used for measuring ridge dimensions) and radiographically on the cone-beam computed tomography (CBCT) and comparing the results of the study group (20 sockets) with the control group (the other 20sockets), to assess the effectiveness of Demineralized Dentin Allograft for ridge preservation

SECONDARY OUTCOMES:
Assess and comparing the mouth opening of both groups | One day post-operative, one week post-operative
  Assess the mouth opening of the patient using a millimeter ruler (by measuring the distance between maxillary incisal edge and mandibular incisal edge) and comparing the results of both groups
Assess and comparing the swelling of both groups | One day post-operative, one week post-operative
  Swelling levels after surgery will be measured using anatomic landmarks (Tragus-Labial commissure and Tragus-Pogonion), the distances between the landmarks used for the evaluation methods will be measured before the operation.
  All measurements will be done using millimeter ruler, while the patient will be seated.
Assess and comparing the pain of both groups | One day post-operative, one week post-operative
  we will use the Visual Analogue Scale (VAS) for pain measurement
Assess and comparing the soft tissue parameters (bleeding on probing and color of the gingiva) of both groups | One day post-operative, one week post-operative
  The bleeding on probing will be assessed by using periodontal probe and this will be done around mandibular first and second molars

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Habib, B.D.S, Principal Investigator — Faculty of Dentistry- Horus University in Egypt; Ahmed Khalil, Study Director — Faculty of Dentistry- Horus University in Egypt; Eman Abdelsalam, Study Director — Faculty of Dentistry- Horus University in Egypt
Locations (1):
- Faculty of Dentistry- Horus University in Egypt, Damietta, New-Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi CP, D'Lima CB, Samat UC, Karde PA, Patil AG, Dani NH. Comparative Alveolar Ridge Preservation Using Allogenous Tooth Graft versus Free-dried Bone Allograft: A Randomized, Controlled, Prospective, Clinical Pilot Study. Contemp Clin Dent. 2017 Apr-Jun;8(2):211-217. doi: 10.4103/ccd.ccd_147_17. PMID 28839405
- [Background] Grover V, Kapoor A, Malhotra R, Sachdeva S. Bone allografts: a review of safety and efficacy. Indian J Dent Res. 2011 May-Jun;22(3):496. doi: 10.4103/0970-9290.87084. PMID 22048602